CLINICAL TRIAL: NCT03448809
Title: A Randomized Feasibility Trial of a New Transdiagnostic Cognitive and Behavioral Intervention Versus Treatment as Usual in School-aged Children With Emotional and Behavioral Disturbances
Brief Title: Randomized Feasibility Trial of Mind My Mind
Acronym: MindMyMind
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: TrygFonden, Denmark (Industry); The Danish Mental Health Foundation (Other)
Responsible Party: Principal Investigator, Pia Jeppesen, Ph.D., Senior Researcher and Specialist in Child and Adolescent Psychiatry, and Associate Professor, Institute for Clinical Medicine, Faculty of Health and Medical Sciences, University of Copenhagen, Denmark, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMMpilotrct
Record Dates: First submitted 2017-11-08; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Anxiety; Anxiety Disorders; Depressive Symptoms; Depressive Disorder; Problem Behavior; Oppositional Defiant Disorder; Conduct Disorder; Behavior Disorders
Keywords: Cognitive and Behavioral Therapies; Children and Adolescents; Community Health Care; Early Intervention; Feasibility Study
MeSH Terms: conditions — Anxiety Disorders; Depression; Depressive Disorder; Problem Behavior; Oppositional Defiant Disorder; Conduct Disorder; Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: No sample size calculation was performed for this parallel, two-arm feasibility RCT. Because the study population was heterogeneous and included children with a broad spectrum of emotional and behavioral mental health problems, 100-120 children were needed in the new experimental MMM arm to answer the research questions related to implementation and acceptability of the MMM manual. Therefore the goal was to include 150 children to be randomly allocated (3:1) to MMM versus TAU. The central, computerized randomization was performed by DEFACTUM using concealed computer-generated allocation sequences with variable block size, and stratification by region (Zealand or Central Denmark), and by age (6-10 years or 11-16 years).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMM (Mind My Mind training) (Experimental): Mind My Mind training
  Interventions: Behavioral: Mind My Mind
- TAU (Treatment as Usual) (Active Comparator): Treatment as Usual
  Interventions: Behavioral: TAU (Treatment as Usual)

INTERVENTIONS:
Behavioral: Mind My Mind — An individual, modular and flexible cognitive and behavioural therapy
  Arms: MMM (Mind My Mind training)
Behavioral: TAU (Treatment as Usual) — The children were offered anonymous counselling, supportive talk therapy, pedagogical advice, network meetings, and/or individual support in the school setting. A few were offered group-based CBT-programs for selected problems, but the access to manualized treatment was generally very restricted.
  Arms: TAU (Treatment as Usual)

SUMMARY:
In this feasibility RCT of the modular and flexible cognitive and behavioural therapy (Mind My Mind, MMM) compared with treatment as usual, the overall research aim was to explore the trial design and the acceptability of the assessments, interventions and outcome measures among children, parents, teachers and therapists, and secondly to provide data to estimate the parameters required to design a definitive RCT.

DETAILED DESCRIPTION:
Background and aims:

Emotional and behavioral disorders are common in youths, and large-scale implementation of evidence-based treatments lack behind the needs of the population. The Mind My Mind (MMM) study in Denmark is a multidisciplinary collaborative effort to adapt current evidence-based treatment strategies for implementation with school children in diverse municipalities in Denmark. The overarching goals of the Mind My Mind study are to develop, implement, evaluate and disseminate a program for the prevention and treatment of children's emotional and behavioral disturbances at the lowest effective level.

Methods:

A parallel, two-arm trial compared the modular and flexible cognitive and behavioral therapy (Mind My Mind, MMM) with treatment as usual (TAU) for children aged 6-16 years with subclinical or clinical levels of emotional and behavioral difficulties.

The trial was conducted in diverse municipalities in Denmark in the period from December 2015 to March 2017. Participants were help-seeking school-children with indicated needs for psychological help. The help-seeking children entered a two-stage screening for eligibility by web-based standardized psychometric instruments: 1) the strengths and difficulties questionnaire (SDQ), 2) the Child Behaviour Checklist (CBCL) and the Youth Self-Report (YSR). This screening procedure was set up as a new routine in the Pedagogical Psychological Services (PPR) in the Municipalities. The screening enabled PPR to identify children with anxiety, depressive symptoms and/or behavioral problems causing distress/impact in their daily life (eligible for the study) versus those with too mild problems (excluded based on SDQ-parent-scores below a pre-specified cut-off according to an algorithm) or too severe problems (excluded and referred to the Child and Adolescent Psychiatry or other specialized services). If the child was eligible, both parents were asked to give informed consent to inclusion of the child in the research study.

The included children were randomized (3:1) to MMM versus TAU. All outcomes were measured by use of self-, parent-, and teacher-reported questionnaires covering specific and general psychopathology, daily and social functioning, quality of life of the child, and parental distress at baseline, week 14 and week 22. At entry, the child and the parent formulated each three problems that they wanted to change. The Top-3-problems were written into the web-based questionnaire using their own words. Then, each problem was scored on a 10-point likert scale along with scoring of the Brief Problem Monitor (BPM) by the child and the parent separately. These scores were collected weekly during the treatment period, at end of treatment (week 14) and at follow-up (week 22). The satisfaction with the MMM sessions was also scored weekly (MMM arm only).

The primary objectives and outcomes measures:

1. To assess the flow of participants through the visitation
2. To explore whether the visitation procedures, and the inclusion and exclusion criteria were applicable and appropriate for the recruitment. The included and the excluded children were described and compared with regard to the family and social characteristics, and the type and severity of psychopathology as measured with the SDQ, CBCL and YSR.
3. To assess the retention of children in the MMM arm.
4. To assess the proportion of children in the MMM arm who were referred to more specialized services during the study period.
5. To assess the satisfaction with MMM sessions among children and parents in the MMM arm.
6. To describe the dosing and sequencing of the MMM modules as reported by the therapists after each session and compare the actual use of the MMM manual with the intended use according to the manual.

The secondary objectives and outcomes measures:

1. To measure the key outcome domains with regard to completion rates, missing data, and the estimated differences between MMM and TAU.
2. To perform an initial validation of the Top-3-problem-scores by studying the correlations between the scores within and across informants, across time, and the correlations between the Top-3-problem-scores and the BPM-scores.

Statistical analyses:

The feasibility measures were summarized using standard descriptive statistics. The group differences in outcome were analyzed in intention-to-treat (ITT) analyses using mixed models repeated measures or linear regression analyses with multiple imputations.

Perspectives:

The new modular and flexible manual, the centralized education and supervision of the psychologists, and the web-based data collection with feedback in real time was implemented in an explanatory feasibility trial to prepare for a future definitive RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6-16 years and in 0-9th grade (excluding the second semester of the 9th grade).
2. Bother genders.
3. Child and/or parents report that the child has problems within the domains of anxiety, depressive symptoms and behavioral problems.
4. SDQ scores reported by the parent are above the lower cutoff: a total difficulties score of ≥14 and/or emotional problems ≥5; combined with a functional impairment score of ≥1.
5. The child and at least one of the two parents understand and speak Danish sufficiently to participate in the treatment.
6. Written informed consent from the holders of the parental rights and responsibilities (usually both parents).

Exclusion Criteria:

1. Indications based on the available information that the child may have a severe mental disorder like autism spectrum disorder, ADHD, schizophrenia-like psychosis, an eating disorder, or other mental disorder requiring referral to a more intensive assessment or treatment in child and adolescent mental health services (after systematic assessment and according to the usual recommendations and guidelines).
2. Indications of intellectual functional impairment, severe learning difficulties or other special needs that would interfere negatively with the MMM training. The judgment is made as a best estimate by the PPR psychologist on the basis of the available information. A formal intelligence test is not required.
3. The child has a clinically significant abuse of alcohol or psychoactive drugs
4. Parents did not answer the SDQ and CBCL during visitation

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2017-04-02 (Actual); Study Completion 2017-04-02 (Actual)

PRIMARY OUTCOMES:
The flow of participants through the visitation. | At baseline (week 0).
  The number of children/parents who accepted the invitation to sign up for visitation to the study The number successfully screened and assessed for eligibility. The number estimated to be eligible. The proportion of eligible children for whom the parents gave informed consent to let the child participate in the research study.
  The number excluded in total, and calculated for each inclusion and exclusion criteria.
The family and social background characteristics. | At baseline (week 0).
  One of the parents served as an informant. The questionnaire was developed for the Mind My Mind and asked about the family composition including if parents are separated, divorced or living together, how much time the child spend with each parent, early developmental problems, physical and mental health problems and disorders, school problems related to learning, social functioning and absence from school, child's history of having received any pedagogical educational support, medicine, psychological or psychiatric treatments; and parents' education and self-reported mental health problems.
The Strengths and Difficulties Questionnaire (SDQ). | At baseline (week 0).
  SDQ contains 25 items, each scored on a 3-point Likert scale (0, 1, 2), and divided into five sub-scales measuring emotional problems, behavioral problems, hyperactivity, peer problems and pro-social behavior. The extended version included questions about child distress and interference of problems with home-life, friendships, classroom learning and leisure activities, summed up the distress and the interference of problems in the impact score (range 0-10).
  For screening purposes, high-risk and low-risk groups were defined by cut-offs for the top 10th percentile of the Danish population. Informants: The SDQ was answered by the child (only age 11 -16 years) and the parent. For those children included in the research trial, the school teacher was requested to answer the SDQ.
The retention of children in the MMM arm. | At end of treatment (week 14).
  The proportion continuing training until the agreed and planned ending (minimum 9 sessions) among the total number of children being allocated to MMM training.
The proportion of children in the MMM arm who were referred to more specialized services during the study period. | At end of treatment (week 14)
  The number referred to child and adolescent psychiatry or other specialized services according to the mandatory records made by the psychologist at end of the each MMM training.
The satisfaction with MMM sessions among children and parents in the MMM arm. | Within one week after each MMM session.
  The questionnaire contains six questions: 1) I liked the last meeting, 2) I learned something new at the last meeting, 3) All in all, I understood the tasks, 4) I can use what I learned at the last meeting, 5) I felt that the trainer understood me, 6) The trainer presented the tasks in a good way for me.
  The questionnaire was scored after each MMM session by the child or by the parent, depending on who was the primary recipient in the given session (as recorded by the therapist). Each question was scored on 5-point likert-scale, score 1 = "very unsatisfied" and 5 = "very satisfied".
The dosing and sequencing of the MMM modules. | Within one day after each MMM session.
  The trainer made a record of each training session including information on the current principal problem domain (anxiety, depressive symptoms, behavioural problems), the selected path, modules and worksheets used in the session, the participant (child, parents) the primary recipient, and, if it was the last session, how the training ended (ending as planned, drop out, referral to support/treatment outside the manual).
The authorized Danish version of the Achenbach System of Empirically Based Assessment (ASEBA), Child Behaviour Checklist (CBCL). | At baseline (week 0)
  The Child Behaviour Checklist for 6-16-year-olds was answered by the parent. The part with 112 problem items was used. These are statements answered on a Likert scale: zero equals "not true", one equals "partly true or sometimes", two equals "very true or frequently". CBCL derives total problem score, and subscale scores for externalizing and internalizing problems.
The authorized Danish version of the Achenbach System of Empirically Based Assessment (ASEBA), the Youth Self-Report (YSR). | At baseline (week 0)
  The YSR was answered by the child (age 11-16- years). The part with 112 problem items was used. These are statements answered on a Likert scale: zero equals "not true", one equals "partly true or sometimes", two equals "very true or frequently". YSR derives total problem score, and subscale scores for externalizing and internalizing problems.

SECONDARY OUTCOMES:
Spence Children's Anxiety Scale (SCAS) | Baseline (week 0), end of treatment (week 14), and follow-up (week 22).
  The SCAS comprises parent- and youth-reported questionnaires with 38 and 44 items, respectively. Each is rated on a four-point scale (0-1-2-3). The self-reported version is longer because it includes six positive filler items. The SCAS consists of six subscales reflecting symptoms specifically related to social phobia (SoP; six items), panic disorder and agoraphobia (Panic; nine items), generalized anxiety disorder (GAD; six items), obsessive-compulsive disorder (OCD; six items), separation anxiety disorder (SAD; six items) and fear of physical injury (Fear; five items). Each subscale is scored separately and added together for a total score reflecting overall anxiety symptoms. A validation of the Danish version of the SCAS in children and adolescents aged 7-17 years found good psychometric properties.
The Mood and Feelings Questionnaire (MFQ) | Baseline (week 0), end of treatment (week 14), and follow-up (week 22).
  The MFQ comprises parent- and youth-reported questionnaires with 34 and 33 items, respectively; each rated on a three-point scale (0-1-2). The MFQ have well-established predictive validity for detection of depressive states and suicidality in epidemiological and clinical samples of children and adolescents aged 8-17 years, and the parent-reported MFQ has also demonstrated sensitivity for change with treatment.
The KIDSCREEN | Baseline (week 0), end of treatment (week 14), and follow-up (week 22).
  The KIDSCREEN is a Health-Related Quality of Life (HRQOL) questionnaire for children and adolescents aged from 8 to 18 years.
  It comprises parent- and youth-reported questionnaires with 27 items, each rated on a five point scale (1-2-3-4-5).
  It contains five dimensions (subscales): Physical Well-Being, Psychological Well-Being, Autonomy & Parents, Peers & Social Support and School Environment.
Eyberg Child Behaviour Inventory (ECBI) | Baseline (week 0), end of treatment (week 14), and follow-up (week 22).
  The ECBI is a brief, parent-reported behavioral rating scale of externalizing problems in children of age 2-16 years. It consists of 36 items that assess typical problem behavior reported by parents of children with oppositional and conduct disorders. Each item is rated on a 7-point Intensity Scale that indicates how often the behaviors currently occur (0=Never, 4=sometimes, 7=always); and a Problem scale that identifies whether the child's behavior is problematic or not for the parent (1=yes, 0=no). Hence, the sum of scores on the Intensity Scale measures the overall intensity with which the child displays the behaviors, while the sum of scores on the Problem scale measures the number of problematic behaviors.
Weiss Functional impairment rating Scale (WFIRS) | Baseline (week 0), end of treatment (week 14), and follow-up (week 22).
  The Weiss Functional Impairment Rating Scale-Parent Report (WFIRS) was designed to evaluate to what degree a child's behavior or emotional problems impacted various domains of daily functioning. It comprises parent- and youth-reported questionnaires with 50 items, each rated on a four-point scale (0-1-2-3). Although it has only been validated (and found very sensitive for change) in clinical samples of children aged 6-17 years with ADHD, it focuses on the impact of emotional and behavioral problems, and hence shows good face validity as a measurement of daily functioning in a much broader group of children with emotional and behavioral problems. The WFIRS covers six dimensions of functioning (subscales): Family and home life, School and learning, Life skills, Self-Concept, Social activities, and Risk behaviors. Only the parent-reported version was used in the present study.
Parental Stress Scale (PSS) | Baseline (week 0), end of treatment (week 14), and follow-up (week 22).
  The PSS comprises a parent-reported questionnaire with 18 items, each rated on a five point scale (0-1-2-3-4). It measures the stress a parent may experience as parent of children and adolescents of age 0-18 years. The PSS is currently being validated in Denmark.
The Experience of Service Questionnaire (ESQ) | Baseline (week 0), end of treatment (week 14), and follow-up (week 22).
  The ESQ comprises parent- and youth-reported questionnaires with 7 items, each rated on a three-point scale (0-1-2). The Danish version was adapted from a longer English questionnaire asking young people and their parents how they felt about the psychiatric service they received. The brief Danish version proved useful in a recent study of the Cool Kids program in the community.
Top-3-problems | Baseline (week 0), weekly during treatment, end of treatment (week 14), and follow-up (week 22).
  As part of the visitation, the child and the parent were asked to separately identify three problems (Top-3-problems) causing distress or otherwise impacting on the daily life of the child.
  The question to the child: "Try to choose the three issues that are most important for you to do something about, because they make you feel uncomfortable or they prevent you from doing the things, you want to do. Please choose which problem is number 1 (the largest), number 2 (second largest) and number 3. We call them your Top-3-problems." The respondent then enter their own formulation of the three "Top-3-problems" into the web-based questionnaire (thereby personalizing the questionnaire), after which they each score each problem on a 10-point scale (0-1-2….10), where a score of 10 means "worst you can imagine", and 1 means "so little that it does not matter at all." The child and the parent each scored their own set of The child and the parent each scored.
The Brief Problem Monitor (BPM) | Baseline (week 0), weekly during treatment, end of treatment (week 14), and follow-up (week 22).
  This standardized questionnaire, BPM, consists of three subscales (internalizing problems, attention problems, externalizing difficulties), and a total problems scale. The 19 items are derived from the CBCL/YSR. The brief scale is designed to monitor children's responses to interventions over periods of days, weeks, or months, and their level of functioning during the course.
  The child and the parent each scored the BPM right after the Top-3-problems.
The Strengths and Difficulties Questionnaire (SDQ). | Baseline (week 0), weekly during treatment, end of treatment (week 14), and follow-up (week 22).
  SDQ contains 25 items, each scored on a 3-point Likert scale (0, 1, 2), and divided into five sub-scales measuring emotional problems, behavioral problems, hyperactivity, peer problems and pro-social behavior. The extended version included questions about child distress and interference of problems with home-life, friendships, classroom learning and leisure activities, summed up the distress and the interference of problems in the impact score (range 0-10).
  For screening purposes, high-risk and low-risk groups were defined by cut-offs for the top 10th percentile of the Danish population. Informants: The SDQ was answered by the child (only age 11 -16 years) and the parent. For those children included in the research trial, the school teacher was requested to answer the SDQ.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jeppesen, Ph.D., Principal Investigator — Child and Adolescent Mental Health Centre, Mental Health Services of the Capital Region of Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James A, Soler A, Weatherall R. Cognitive behavioural therapy for anxiety disorders in children and adolescents. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD004690. doi: 10.1002/14651858.CD004690.pub2. PMID 16235374
- [Background] Reynolds S, Wilson C, Austin J, Hooper L. Effects of psychotherapy for anxiety in children and adolescents: a meta-analytic review. Clin Psychol Rev. 2012 Jun;32(4):251-62. doi: 10.1016/j.cpr.2012.01.005. Epub 2012 Feb 13. PMID 22459788
- [Background] Merry SN, Hetrick SE, Cox GR, Brudevold-Iversen T, Bir JJ, McDowell H. Psychological and educational interventions for preventing depression in children and adolescents. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD003380. doi: 10.1002/14651858.CD003380.pub3. PMID 22161377
- [Background] Stice E, Shaw H, Bohon C, Marti CN, Rohde P. A meta-analytic review of depression prevention programs for children and adolescents: factors that predict magnitude of intervention effects. J Consult Clin Psychol. 2009 Jun;77(3):486-503. doi: 10.1037/a0015168. PMID 19485590
- [Background] Weisz JR, McCarty CA, Valeri SM. Effects of psychotherapy for depression in children and adolescents: a meta-analysis. Psychol Bull. 2006 Jan;132(1):132-49. doi: 10.1037/0033-2909.132.1.132. PMID 16435960
- [Background] Furlong M, McGilloway S, Bywater T, Hutchings J, Smith SM, Donnelly M. Behavioural and cognitive-behavioural group-based parenting programmes for early-onset conduct problems in children aged 3 to 12 years. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD008225. doi: 10.1002/14651858.CD008225.pub2. PMID 22336837
- [Background] Mytton J, DiGuiseppi C, Gough D, Taylor R, Logan S. School-based secondary prevention programmes for preventing violence. Cochrane Database Syst Rev. 2006 Jul 19;2006(3):CD004606. doi: 10.1002/14651858.CD004606.pub2. PMID 16856051
- [Background] McCarty DL, Surpure JS. Emergency management of the acutely poisoned child/adolescent. Indian J Pediatr. 1990 Mar-Apr;57(2):223-34. doi: 10.1007/BF02722093. No abstract available. PMID 2246021
- [Background] Wilson SJ, Lipsey MW. School-based interventions for aggressive and disruptive behavior: update of a meta-analysis. Am J Prev Med. 2007 Aug;33(2 Suppl):S130-43. doi: 10.1016/j.amepre.2007.04.011. PMID 17675014
- [Background] Stoltz S. Stay Cool Kids?! Effectiveness, Moderation and Mediation of a Preventive Intervention for Externalizing Behavior. Utrecht University Repository (2012).
- [Background] Bilenberg N. The Child Behavior Checklist (CBCL) and related material: standardization and validation in Danish population based and clinically based samples. Acta Psychiatr Scand Suppl. 1999;398:2-52. doi: 10.1111/j.1600-0447.1999.tb10703.x. PMID 10687023
- [Background] Bordin IA, Rocha MM, Paula CS, Teixeira MC, Achenbach TM, Rescorla LA, Silvares EF. Child Behavior Checklist (CBCL),Youth Self-Report (YSR) and Teacher's Report Form(TRF): an overview of the development of the original and Brazilian versions. Cad Saude Publica. 2013 Jan;29(1):13-28. doi: 10.1590/s0102-311x2013000100004. PMID 23370021
- [Background] Rescorla LA, Ginzburg S, Achenbach TM, Ivanova MY, Almqvist F, Begovac I, Bilenberg N, Bird H, Chahed M, Dobrean A, Dopfner M, Erol N, Hannesdottir H, Kanbayashi Y, Lambert MC, Leung PW, Minaei A, Novik TS, Oh KJ, Petot D, Petot JM, Pomalima R, Rudan V, Sawyer M, Simsek Z, Steinhausen HC, Valverde J, Ende Jv, Weintraub S, Metzke CW, Wolanczyk T, Zhang EY, Zukauskiene R, Verhulst FC. Cross-informant agreement between parent-reported and adolescent self-reported problems in 25 societies. J Clin Child Adolesc Psychol. 2013;42(2):262-73. doi: 10.1080/15374416.2012.717870. Epub 2012 Sep 25. PMID 23009025
- [Background] Goodman A, Goodman R. Strengths and difficulties questionnaire as a dimensional measure of child mental health. J Am Acad Child Adolesc Psychiatry. 2009 Apr;48(4):400-403. doi: 10.1097/CHI.0b013e3181985068. PMID 19242383
- [Background] Goodman R, Meltzer H, Bailey V. The Strengths and Difficulties Questionnaire: a pilot study on the validity of the self-report version. Eur Child Adolesc Psychiatry. 1998 Sep;7(3):125-30. doi: 10.1007/s007870050057. PMID 9826298
- [Background] Goodman R. The extended version of the Strengths and Difficulties Questionnaire as a guide to child psychiatric caseness and consequent burden. J Child Psychol Psychiatry. 1999 Jul;40(5):791-9. PMID 10433412
- [Background] Daviss WB, Birmaher B, Melhem NA, Axelson DA, Michaels SM, Brent DA. Criterion validity of the Mood and Feelings Questionnaire for depressive episodes in clinic and non-clinic subjects. J Child Psychol Psychiatry. 2006 Sep;47(9):927-34. doi: 10.1111/j.1469-7610.2006.01646.x. PMID 16930387
- [Background] Arendt K, Hougaard E, Thastum M. Psychometric properties of the child and parent versions of Spence children's anxiety scale in a Danish community and clinical sample. J Anxiety Disord. 2014 Dec;28(8):947-56. doi: 10.1016/j.janxdis.2014.09.021. Epub 2014 Oct 16. PMID 25445085
- [Background] Reedtz C, Bertelsen B, Lurie J, Handegard BH, Clifford G, Morch WT. Eyberg Child Behavior Inventory (ECBI): Norwegian norms to identify conduct problems in children. Scand J Psychol. 2008 Feb;49(1):31-8. doi: 10.1111/j.1467-9450.2007.00621.x. PMID 18190400
- [Background] Burns GL, Patterson DR. Factor structure of the Eyberg Child Behavior Inventory: a parent rating scale of Oppositional Defiant Behavior Toward Adults, Inattentive Behavior, and Conduct Problem Behavior. J Clin Child Psychol. 2000 Dec;29(4):569-77. doi: 10.1207/S15374424JCCP2904_9. PMID 11126634
- [Background] Ravens-Sieberer U, Auquier P, Erhart M, Gosch A, Rajmil L, Bruil J, Power M, Duer W, Cloetta B, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J; European KIDSCREEN Group. The KIDSCREEN-27 quality of life measure for children and adolescents: psychometric results from a cross-cultural survey in 13 European countries. Qual Life Res. 2007 Oct;16(8):1347-56. doi: 10.1007/s11136-007-9240-2. Epub 2007 Aug 1. PMID 17668292
- [Background] Tarakcioglu MC, Memik NC, Olgun NN, Aydemir O, Weiss MD. Turkish validity and reliability study of the Weiss Functional Impairment Rating Scale-Parent Report. Atten Defic Hyperact Disord. 2015 Jun;7(2):129-39. doi: 10.1007/s12402-014-0158-6. Epub 2014 Nov 27. PMID 25428590
- [Background] Oronoz B, Alonso-Arbiol I, Balluerka N. A Spanish adaptation of the Parental Stress Scale. Psicothema. 2007 Nov;19(4):687-92. PMID 17959127
- [Background] Attride-Stirling J, Humphrey C, Tennison B, Cornwell J. Gathering data for health care regulation: learning from experience in England and Wales. J Health Serv Res Policy. 2006 Oct;11(4):202-10. doi: 10.1258/135581906778476607. PMID 17018193